CLINICAL TRIAL: NCT01583140
Title: Culturally and Linguistically Adapted Physical Activity Intervention for Latinas (Seamos Saludables)
Brief Title: Seamos Saludables - Physical Activity Intervention Study for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Dr.Bess Marcus, Professor and Chair, Department of Family and Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SALUDABLES-2009; 5R01NR011295 (NIH)
Record Dates: First submitted 2012-03-06; First posted 2012-04-23 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; Latinas
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention (Experimental): Culturally-modified, individually tailored physical activity print materials
  Interventions: Behavioral: Physical Activity Intervention
- Control (Active Comparator): Bilingual health education booklets
  Interventions: Behavioral: Wellness control

INTERVENTIONS:
Behavioral: Wellness control — Participants in the Wellness Control arm of the study receive a variety of print materials focused on general health topics.
  Arms: Control
Behavioral: Physical Activity Intervention — Participants in the Physical Activity Intervention arm of the study receive culturally-modified, individually tailored physical activity print materials.
  Arms: Exercise Intervention

SUMMARY:
In this study the investigators are specifically targeting Latina women because they are more likely to be inactive and, therefore, are at higher risk for developing chronic conditions like obesity, diabetes, or cardiovascular disease. Through focus groups and cognitive interviews with Latinas in the Providence area, the investigators have modified our print-based intervention, already tested and proven to be effective in English-speaking communities, to be culturally and linguistically appropriate for the Latina community.

The objective of Seamos Saludables is to determine whether this culturally tailored print intervention will produce greater increases in physical activity levels among Latina women than a program focused on general health topics. Participants are randomly assigned to one of two groups (exercise and general wellness) and attend 4 clinic visits to complete baseline and follow-up assessments.

The investigators hypothesize that at the end of treatment, intervention participants will report significantly more minutes of at least moderate intensity physical activity per week than the wellness contact control participants.

DETAILED DESCRIPTION:
In the U.S., Latinos report higher rates of inactivity and related health conditions (e.g., hypertension,hypercholesteremia, obesity, heart disease, stroke, diabetes) than non-Hispanic whites. Furthermore, Latino women (Latinas) report higher rates of sedentary behavior than Latino men. Due to cultural factors, socioeconomic circumstances, differences in educational background, and language barriers, Latinos in general, and especially Latinas, have limited access to public health interventions that promote physically active lifestyles. To address this public health crisis, effective interventions that leverage state-of-the-art theory and methods are needed. The investigators research group has 20 years experience developing and evaluating individually tailored computer expert system-driven physical activity interventions (based on Social Cognitive Theory and the Transtheoretical Model). In the investigators recent pilot study (R21NR009864), the investigators culturally and linguistically adapted the existing tailored intervention for sedentary Latinas and conducted a small randomized trial of the modified program (N=94). Six month (post-intervention) assessments are still ongoing, but three month data have been collected on 87 participants (93% retention). Intervention participants increased their physical activity from a mean of 17 minutes per week (SD=25.8) at baseline to 92 minutes (SD=69.8) at three months, whereas contact control participants reported increasing their physical activity from 12 minutes per week (SD=21.8) at baseline to 64 minutes (SD=84.3) at three months. The trends in the means at 3 months lend preliminary support for the efficacy of the intervention and the high retention rates, especially for a study targeting a hard-to-reach group like Latinas, bode well for its feasibility and acceptability. For the current proposal, the investigators will build on these encouraging results by conducting an adequately powered (N=312) randomized controlled trial to test the efficacy of the culturally and linguistically modified, individually tailored print intervention compared with a wellness contact control condition (e.g., cardiovascular health information from NHLBI in Spanish). Data will be collected at baseline, 6, and 12 months using well-established physical activity measures (7-Day PAR, Actigraphs), as well as a comprehensive set of psychosocial questionnaires. The investigators hypothesize that at the end of treatment, intervention participants will report significantly more minutes of at least moderate intensity physical activity per week than the wellness contact control participants. The investigators will also examine the maintenance of treatment effects at 12 months, costs of delivering the tailored intervention program, and potential mediators and moderators of the intervention-physical activity relationship. In the proposed study the investigators seek to promote physical activity among this at-risk population using a high-reach, low-cost strategy, which has great potential for adoption on a larger scale and thus high potential for reducing existing health disparities in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Generally healthy
* Sedentary (Less than 60 minutes per week of mod or vigorous physical activity)
* Latina (self-defined)
* Must be able to read and write Spanish fluently
* 18 - 65 years of age
* Planning on living in the area for the next 12 months

Exclusion Criteria:

* Pregnant or planning on becoming pregnant
* BMI greater than 45
* Not able to walk continuously for 30 minutes/limited ability to complete daily activity or ability to exercise
* Exercise is against advice of doctor
* Heart disease/treatment
* Heart murmur
* Angina/chest pain or Angina/chest pain with exertion
* Palpitations
* Stroke/TIA
* Peripheral vascular disease
* Diabetes I or II
* Chronic Infectious Disease - HIV, Hepatitis
* Chronic liver disease
* Cystic fibrosis
* Abnormal EKG on last EKG performed
* Emphysema, Chronic bronchitis, COPD
* Seizure in past year
* Surgery in past year on heart, lung, joint, orthopedic surgery
* Surgery pending in next year on lung, joint, orthopedic surgery
* Unusual/concerning shortness of breath
* Asthma
* High blood pressure/high blood pressure medication
* Abnormal medical Stress Test
* musculoskeletal problems
* Fainting/dizziness more than 3 times in past year OR interferes with daily activities OR causes loss of balance
* Cancer treatment in past 3 months
* Hospitalized for psychiatric disorder in past 3 years or suicidal
* 3 or more alcoholic beverages 5 or more days per week

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in total weekly minutes of physical activity as measured by the 7-Day PAR (Physical Activity Recall), from Baseline to 6-months and 12-months | 6 and 12 months
  The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities including time spent sleeping and in moderate, hard, and very hard activity. The 7-Day PAR is used across many studies in physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other more objective measures of activity levels, along with sensitivity to changes in both moderate and intensive levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- Brown University Institute for Community Health Promotion, Providence, Rhode Island, United States

REFERENCES:
- [Background] Pekmezi DW, Neighbors CJ, Lee CS, Gans KM, Bock BC, Morrow KM, Marquez B, Dunsiger S, Marcus BH. A culturally adapted physical activity intervention for Latinas: a randomized controlled trial. Am J Prev Med. 2009 Dec;37(6):495-500. doi: 10.1016/j.amepre.2009.08.023. PMID 19944914
- [Derived] Benitez TJ, Dunsiger S, Marquez B, Larsen B, Pekmezi D, Marcus BH. Increases in Muscle-Strengthening Activities Among Latinas in Seamos Saludables. Health Educ Behav. 2022 Jun;49(3):446-454. doi: 10.1177/10901981221074908. Epub 2022 Feb 28. PMID 35227112
- [Derived] Larsen B, Gilmer T, Pekmezi D, Napolitano MA, Marcus BH. Cost effectiveness of a mail-delivered individually tailored physical activity intervention for Latinas vs. a mailed contact control. Int J Behav Nutr Phys Act. 2015 Nov 11;12:140. doi: 10.1186/s12966-015-0302-5. PMID 26559336
- [Derived] Marcus BH, Dunsiger SI, Pekmezi D, Larsen BA, Marquez B, Bock BC, Gans KM, Morrow KM, Tilkemeier P. Twelve-month physical activity outcomes in Latinas in the Seamos Saludables trial. Am J Prev Med. 2015 Feb;48(2):179-182. doi: 10.1016/j.amepre.2014.08.032. Epub 2014 Nov 6. PMID 25442225